CLINICAL TRIAL: NCT05107934
Title: International, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of RPH-104 Treatment in Patients With Recurrent Pericarditis
Brief Title: Efficacy and Safety of RPH-104 Treatment in Patients With Recurrent Pericarditis
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: due to the decision of company Top management. No subjects were recruited, none of sites were initiated
Sponsor: R-Pharm Overseas, Inc. (Industry)
Collaborators: Data Management 365 (Industry); Keystat, LLC (Industry)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CL04018106
Record Dates: First submitted 2021-10-28; First posted 2021-11-04 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Recurrent Pericarditis
Keywords: RPH-104; subcutaneous
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RPH-104 80 mg (Experimental): Patients will receive RPH-104 dose 160 mg subcutaneously on Day 0, and 80 mg on Day 7, Day 14 and thereafter once in two weeks.
  Interventions: Biological: RPH-104
- Placebo (Placebo Comparator): Patients (who achieved clinical response defined above by the randomized withdrawal baseline) will receive placebo subcutaneously once every 2 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: RPH-104 — solution for subcutaneous injection, 40 mg/mL
  Arms: RPH-104 80 mg
Drug: Placebo — 0.9% Sodium Chloride solution for Injection
  Arms: Placebo

SUMMARY:
The primary purpose of this study is the evaluation of the efficacy and safety of RPH-104 treatment in patients with recurrent pericarditis.

Pharmacokinetic and pharmacodynamic parameters of RPH-104 multiple doses in this patient population will be assessed as well.

DETAILED DESCRIPTION:
This is a phase 2/3 seamless design study with one interim efficacy analysis. At stage 1 (assuming possible 10% dropout rate in run-in period and screening), around 25 patients will be enrolled. At least 20 patients will be randomized to receive either RPH-104 treatment or placebo.

During the interim analysis, the enrollment won't be paused. Based on interim analysis results the study could be continued or closed. In the case of study continuation, the final estimated sample size is at least 72 patients to be randomized in the withdrawal period (including 20 or more patients randomized in the Stage 1 of the study). Assuming possible 10% dropout in run-in period and 45% dropout in screening period, approximately enrollment of 80 subjects are planned and around 146 subjects will be screened in this study.

The study will consists of five following periods:

1. Screening period (up to 4 weeks). The patients' eligibility for the study will be evaluated based on the eligibility criteria.
2. Run-in (RI) single-blind treatment period (16 weeks) will include single- blind treatment with RPH-104 at a dose 160 mg subcutaneous (SC) on Day 0, and 80 mg on Day 7, Day 14 and thereafter once in two weeks (Q2W) for all patients.

   The RI period includes:
   * 2-weeks Stabilization period, during which blinded RPH-104 is administered on top of standard of care (SOC) pericarditis therapy, and the ongoing pericarditis episode is treated.
   * 10- week Weaning period, during which patients are gradually tapered and stopped background SOC pericarditis therapy, while treatment with blinded RPH-104 continues. corticosteroids (CS) and analgesics (opioid and non-opioid) dose will be tapered starting at RI week 2 and will be stopped by Week 12. NSAIDs and colchicine will be tapered starting at RI Week 6 and will be stopped by Week 12. Opioid analgesics can be continued after Week 12 at stable doses through the end of the OL period if cannot be discontinued without withdrawal symptoms.
   * 4-week Monotherapy period: patients who stopped of background SOC pericarditis therapy will continue to receive blinded RPH-104.

   Patients who discontinue SOC therapy and achieve clinical response at Week 16 are eligible for randomization in the randomized withdrawal (RW) period.
3. Randomized withdrawal (RW) period (24 weeks) includes double-blind treatment with RPH-104 80 mg or placebo Q2W depending on the randomization group.
4. Open-label treatment period (OL) (12 weeks). After completion of the RW period, all subjects that did not discontinue study drug will be transferred to Open-Label (OL) period and will receive open-label RPH-104 80 mg once in two weeks.
5. Safety follow-up period includes monitoring of safety for 8 weeks after the last dosing of the study drug for patients who decided not to participate in open label extension long-term safety study (CL04018108).

The total maximal duration of the study for an individual subject will be approximately 64 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed and dated Informed Consent Form for participation in the study.
* Recurrent pericarditis diagnosis.
* ≥ 1 pericarditis episodes experienced prior to screening has met ≥ 2 of the following 4 criteria, in the Investigator's opinion and based on the documented available data, according to 2015 European Society of Cardiology (ESC) Guidelines for the Diagnosis and Management of Pericardial Diseases:

  * Pericarditic chest pain
  * Pericardial rub
  * New widespread ST-segment elevation/PR-segment depression according to ECG findings
  * Pericardial effusion (new or worsening)
* Presents with at least the third episode of pericarditis during screening (i.e., at least the second pericarditis recurrence following the first pericarditis episode), and within ≤ 7 days prior to and including RI baseline (first administration of study drug) has at least two of the following signs: 1) ≥ 1 day with NRS pain score ≥ 4 (without any other potential causes for the increase in the pain intensity); 2) CRP ≥ 1 mg/dL, (without any other potential causes for the CRP elevation); 3) new or progression of existing pericardial effusion during the diastole as demonstrated by echocardiography; 4) evidence of new widespread ST-elevation (ST segment or T wave ratio in lead v6 > 0.25) or PR depression on ECG. Each sign must be presented either on the same day or separated by no more than 7 days from the other sign.
* NSAIDs and/or colchicine and/or CS (in any combination), if used, at stable dose levels for at least 3 days prior to and including RI baseline before RPH-104 administration.
* If using NSAIDs and/ or colchicine and/or CS at RI baseline, is willing and able, in the opinion of the investigator, to taper and discontinue these drugs no later than Week 12 of the RI period.
* The patient's ability and willingness (in the reasonable opinion of the Investigator) to come to the study site for all scheduled visits, to undergo all study procedures and comply with the protocol requirements, including consent to subcutaneous injections by qualified personnel of the study site.
* Consent of women of childbearing potential (defined as all women physiologically able to become pregnant) to use highly effective contraceptive methods throughout the study, starting from the beginning of the screening (signing of the Informed Consent Form) and for at least 8 weeks after discontinuation of the study drug; and a negative pregnancy test result (serum test for chorionic gonadotropin).

OR

Consent of sexually active male subjects to use highly effective contraceptive methods throughout the study, starting from the beginning of the screening and for at least 8 weeks after discontinuation of the study drug.

Highly effective methods of contraception include the following:

1. complete abstinence (if it agrees with the preferable and usual lifestyle of the patient). [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception];
2. sterilization: bilateral removal of the ovaries (with or without removal of the uterus) or tubal ligation at least 6 weeks before the start of the study therapy. If only the ovaries have been removed, the reproductive status of the woman should be confirmed by subsequent hormone tests;
3. sterilization of the male partner at least 6 weeks before the start of the study therapy (with proper documentation of the absence of sperm cells in the ejaculate after vasectomy) [in female subjects, the sexual partner after vasectomy should be the only partner];
4. use of a combination of any two of the following (a+b or a+c, or b+c):

   1. the use of oral, injectable or implanted hormonal contraceptives; in the case of oral contraceptives, women should consistently use the same drug for a minimum of 3 months prior to the initiation of the study treatment;
   2. placement of an intrauterine device (IUD) or intrauterine system (IUS);
   3. barrier methods of contraception: a condom or occlusive cap (diaphragm or cervical/vault caps) and spermicidal foam/gel/film/cream/vaginal suppository.

      Exclusion Criteria:
      * Hypersensitivity to the study drug (RPH-104), and/or its components/excipients
      * History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies or fusion proteins.
      * Pericarditis secondary to: a) tuberculosis (TB); b) postthoracic blunt trauma; c) myocarditis; d) systemic autoimmune diseases (systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis, etc.; Still's disease and familial Mediterranean fever are not considered as autoimmune diseases); e) neoplastic, purulent, or radiation etiologies.
      * Is currently receiving CS at a dose of > 60 mg/day prednisone (or equivalent).
      * Prior therapy with:

        * rilonacept - less than 6 weeks prior to the baseline assessment (Day 0 of run-in treatment period);
        * canakinumab - less than 12 weeks prior to the baseline assessment (Day 0 of run-in treatment period);
        * anakinra - less than 5 days prior to the baseline assessment (Day 0 of run-in treatment period);
        * Tumor necrosis factor (TNF) inhibitors, Interleukin 6 (IL-6) inhibitors, Janus kinase inhibitors - less than 12 weeks prior to the baseline assessment (Day 0 of run-in treatment period);
        * immunosuppressive agents (azathioprine, cyclosporine, mycophenolate, mofetil, tacrolimus, sirolimus, mercaptopurine) - within 24 weeks prior to the baseline assessment (Day 0 of run-in treatment period), methotrexate - less than two weeks prior to the baseline assessment (Day 0 of run-in treatment period),
        * any other biological preparations less than 5 half-lives prior to the treatment initiation (Day 0 of run-in treatment period).
      * The use of a live (attenuated) vaccine within 3 months prior to Day 0 of the RI treatment period and/or the need to use this type of a vaccine within 3 months after the discontinuation of the study drug. Live attenuated vaccines include vaccines against viral infections such as measles, rubella, mumps, chickenpox, rotavirus, influenza (in the form of a nasal spray), yellow fever, polio (oral polio vaccine); vaccines against tuberculosis (BCG), typhoid (oral typhoid vaccine) and typhus (epidemic typhoid vaccine) vaccines. Patient's immunocompetent family members should refrain from administration of a polio vaccine during the patient's participation in the study.
      * Conditions or signs that, according to the Investigator, indicate impairment (weakening) of the immune response in the patient and/or significantly increase the risk of the use of immunosuppressive therapy, including, but not limited to, the following conditions at the screening:

        * active bacterial, fungal, viral (including COVID-19) or protozoal infection;
        * opportunistic infections and/or Kaposi's sarcoma;
        * chronic bacterial, fungal or viral infection requiring systemic antimicrobial therapy;
        * HIV-infection, hepatitis B or C (patients with treated hepatitis C and negative Polymerase chain reaction (PCR) tests after 3 and 6 months are regarded as cured from hepatitis C and can be included in this study); within 6 months prior to the beginning of the screening period:
        * disseminated herpes zoster infection, herpetic encephalitis, meningitis and other non-self-limiting infections caused by herpes viruses;
      * A history of active tuberculosis or the presence of risk factors or signs indicating the presence of active or latent infection caused by M. tuberculosis, including but not limited to, the following:

        * living in specific conditions that increase the risk of contacts with tuberculosis-infected patients, such as prisoners, gathering of homeless people etc. within a year before the beginning of the screening period;
        * work experience in a healthcare setting with unprotected contacts with patients having high risk of tuberculosis or patients with tuberculosis within a year prior to the beginning of the screening period;
        * close contact, i.e. being in the same room (at home or in another confined environment) for an extended period of time (days or weeks rather than minutes or hours) with a person with active pulmonary tuberculosis within a year prior to the beginning of the screening period;
        * test results indicating active tuberculosis or latent infection caused by M. tuberculosis: positive result of QuantiFERON-TB/T-SPOT test.TB during the screening period; findings of chest X-ray exam in two views confirming pulmonary tuberculosis during the screening period.
      * The presence of any other significant comorbidities (cardiovascular, nervous, endocrine, urinary tract, gastrointestinal tract, liver, blood clotting disorders, autoimmune diseases, etc.) or conditions that may, in the reasonable opinion of the Investigator, adversely affect the participation and well-being of the study subject and/or distort the evaluation of the study results.
      * Uncontrolled diabetes mellitus.
      * History of organ transplant, or the need for transplant surgery at the beginning of the screening period, or elective transplant surgery during the study.
      * The presence of any malignancies during the screening period or within 5 years prior to its initiation, except for non-metastatic basal cell and squamous cell skin cancer after complete resection or carcinoma in situ of any type following complete resection.
      * Mental disorders that, in the reasonable opinion of the Investigator, may affect the patient's participation in the study or his/her ability to comply with the Protocol procedures.
      * Pregnancy or breast-feeding.
      * History of abuse of alcohol or psychoactive substances as assessed by the Investigator.
      * Severe renal impairment (creatinine clearance by Cockcroft-Gault formula <30 mL/min at screening.
      * Presence of any of the following laboratory abnormalities at screening:

        * Absolute neutrophil count <1.5 х 10^9/L,
        * White blood cells (WBC) count <3 х 10^9/L,
        * Platelet count <100 х 10^9/L,
        * Hemoglobin ≤ 80 g/L,
        * Glycated hemoglobin (HbA1c) ≥ 8%,
        * Alanine transaminase (ALT) and/or Aspartate aminotransferase (AST) ≥ 3.0 х Upper limit of normal (ULN),
        * Total bilirubin >1.5 х ULN (except for cases of documented Gilbert's syndrome).
      * Concomitant participation in other clinical studies at the beginning of the screening or the use of any unapproved (investigational) medicinal products within 4 weeks or 5 half-life periods (whichever is longer) up to the baseline assessment (Day 0 of the run-in treatment period).
      * Prior participation in this clinical study (if at least one dose of the study drug was administered). Subjects that are deemed not eligible can be rescreened at the discretion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Time (days) to the pericarditis recurrence within 24 weeks after randomization in patients with recurrent pericarditis treated with RPH-104 compared to placebo. | up to Week 24 (of the RW period)
  Pericarditis recurrence is defined as the occurrence of at least two of the following signs:
  * at least 1 day of pericarditis pain ≥ 4 (on the 11 point numerical rating scale (NRS)) (without any other potential causes for the increase in the pain intensity);
  * at least one CRP value ≥ 1 mg/dL (without any other potential causes for the C-reactive protein (CRP elevation));
  * new or progression of existing pericardial effusion during the diastole as demonstrated by echocardiography;
  * evidence of new widespread ST-elevation (ST segment / T wave ratio in lead v6 > 0.25) or PR depression on electrocardiogram (ECG).
  Each sign can occur either on the same day or separated by no more than 7 days from another sign.

SECONDARY OUTCOMES:
Proportion of subjects who maintained Clinical Response at Week 16 of the RW period in RPH-104 group compared to placebo. | up to Week 16 (of the RW period)
  Clinical response is defined as a weekly average of daily pericarditis pain on the 11-point NRS ≤ 2 AND CRP level ≤ 0.5 mg/dL, AND absent or mild (<10 mm) pericardial effusion during the diastole as demonstrated by echocardiography AND absence of new widespread ST-elevation (ST-segment / T-wave ratio in lead v6 < 0.25), absence of PR depression on ECG AND on monotherapy of randomized study drug at Week 16. (Subjects who had recurrence, discontinued double-blinded treatment, lost to follow-up, and used rescue unblinded RPH-104 or rescue medications (ORT or CSs) before Week 16 will be considered as non-responders.)
Percentage of days with no or minimal pain in the first 16 weeks of the RW period in RPH-104 group compared to placebo. | up to Week 16 (of the RW period)
  No or minimal pain is defined as non-missing NRS ≤ 2.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Lavrovsky, Study Director — R-Pharm Overseas, Inc.
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No